CLINICAL TRIAL: NCT05014789
Title: A Control-IQ Technology 2.0 Feasibility Study in Adult and Adolescent Subjects
Brief Title: Control-IQ Technology 2.0 Adult and Adolescent Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G210146
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes; Control-IQ Technology; automated insulin dosing; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Single arm, Single Center, Prospective Clinical Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Control-IQ 2.0 technology 2.0 on the t:slim X2 insulin pump (Experimental): Each subject will use different combinations of new features of the system each week, in random order, over the next 4 weeks, using the t:slim X2 insulin pump with Control-IQ technology 2.0.
  The first 5 subjects in the study will complete a 48 hour session with multiple challenges during use of Control-IQ technology 2.0, before moving on the outpatient portion of the trial.
  Interventions: Device: Control-IQ technology 2.0

INTERVENTIONS:
Device: Control-IQ technology 2.0 — All subjects wearing the t:slim X2 insulin pump with Control-IQ technology 2.0, and wearing the Dexcom G6 sensor

SUMMARY:
The purpose of this study is to obtain preliminary safety and performance data on planned improvements to Control-IQ technology.

DETAILED DESCRIPTION:
This feasibility study is a prospective, single arm, single center study with a run-in phase, followed by a 48-hour supervised phase, followed by a 4-week at home study with sequential interventions (new feature use). Approximately 30 subjects, both male and female, aged 14 and up, will participate in the study, using new features each week with the t:slim X2 insulin pump with Control-IQ technology.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent male and female subjects >age 14 years
* Clinical diagnosis of Type 1 diabetes for at least one year
* Experienced Control-IQ technology user for ≥3 months.
* Use of Control-IQ technology in closed-loop at least 80% of the 2-week time period before screening.
* Not pregnant or planning a pregnancy during the time period of the study
* Using only Humalog U-100 or Novolog U-100 insulin
* ICR and ISF optimized per investigator judgement
* CGM time in range (70-180 mg/dL) at least 50% on Control-IQ technology
* Has current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (will provide prescription if they do not have one)
* Willing to:

  1. Share Dexcom G6 CGM data with study staff and Tandem
  2. Share t:connect data with Tandem
  3. Eat meals with known carbohydrate amounts
  4. Take meal boluses as directed (use of different options as scheduled and instructed)
  5. Follow study Glycemic Treatment Guidelines for hypo and hyperglycemia
  6. Keep food and exercise diary
  7. Set accurate sleep schedule on pump
  8. Exercise while using exercise activity in Control-IQ technology at least twice weekly
  9. Complete questionnaires before and after using investigational device
  10. Sign an informed consent form
* Willingness to use the Dexcom G6 app on their personal phone throughout the study, and share real time CGM information with a local contact and study staff
* Availability of a local contact who has access to the study participant, knows their whereabouts, and agrees to be promptly available if contacted by study staff. If the subject lives alone, the local contact must live within 30 minutes and have access to the subject overnight.

Exclusion Criteria:

* Diabetic ketoacidosis (DKA) in the past 6 months
* Severe hypoglycemia (needing assistance) in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* History of drug abuse (defined as any illicit drug use) or history of alcohol abuse prior to screening or is unwilling to agree to abstain from illicit drugs throughout the study
* History of heart, lung or kidney disease determined by the investigator to interfere with the study
* Use of glucocorticoids, beta blockers or other medications determined by investigator to interfere with the study
* Use of long-acting insulin or any non-insulin glucose lowering agents (i.e. SGLT-2 inhibitor) other than metformin
* Use of Afrezza during the study period
* Febrile illness within 3 days of the start of the study
* Subject is pregnant or lactating or intending to become pregnant before or during participation in this study
* For subjects >50 years old or with diabetes duration >20 years who will be exercising as part of the 48 hour study, abnormal electrocardiogram consistent with increased risk of arrhythmia, ischemia, or prolonged QTc interval (> 450 ms)
* Significant chronic kidney disease (eGFR < 60) or hemodialysis
* Significant liver disease
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Significant Hypoglycemia | 8 weeks
  CGM percent time <54 mg/dL during each week of feature use, as well as during baseline and run-in periods
Severe hypoglycemia (needing assistance) | 8 weeks
  Number of severe hypoglycemic events (per protocol) during each week of feature use, as well as during baseline and run-in periods
Diabetic Ketoacidosis | 8 weeks
  Number of participants with Diabetic Ketoacidosis (per protocol) during each week of feature use, as well as during baseline and run-in periods
Serious Adverse Events | 8 weeks
  Number of Serious Adverse Events during each week of feature use, as well as during baseline and run-in periods

SECONDARY OUTCOMES:
Percent of time <70 mg/dL | 8 weeks
  CGM percent time <70 mg/dL during each week of feature use, as well as during baseline and run-in periods
Percent of time > 250 mg/dL | 8 weeks
  CGM percent time > 250 mg/dL during each week of feature use, as well as during baseline and run-in periods
Percent of time 70-180 mg/dL | 8 weeks
  CGM percent time in range 70-180 mg/dL during each week of feature use, as well as during baseline and run-in periods
Percent of time 70-140 mg/dL | 8 weeks
  CGM percent time in range 70-140 mg/dL, during each week of feature use, as well as during baseline and run-in periods
Postprandial glycemic peak mg/dL | 8 weeks
  Peak CGM glucose after each meal, during each week of feature use, as well as during baseline and run-in periods
CGM Metrics by time of day | 8 weeks
  Calculate all CGM metrics listed above (including the primary outcome) for: All 24 hours of the day, Daytime only, and Nighttime only.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E Pinsker, MD, Study Chair — Tandem Diabetes Care, Inc.
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No